CLINICAL TRIAL: NCT03145675
Title: Optimizing the Anticoagulation Regimen of Enoxaparin During Percutaneous Coronary Intervention
Brief Title: Optimizing the Anticoagulation Regimen of Enoxaparin During Percutaneous Coronary Intervention (OPTIENOX-PCI)
Acronym: OPTIENOX-PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LiuZhenyu, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-2016-2.24; JS-1286 (Other: Ethics Committee of Peking Union Medical College Hospital)
Record Dates: First submitted 2017-04-14; First posted 2017-05-09 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Anticoagulation; Enoxaparin; Dose
MeSH Terms: conditions — Coronary Artery Disease | interventions — Enoxaparin; Population Groups

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomly assigned into the Planned Staged-dose Group and the Planned Single-dose Group.
  All patients in the Planned Staged-dose Group will receive enoxaparin 0.5 mg/kg at the beginning of coronary angiography. Those with definite indication for subsequent PCI will be given additional enoxaparin 0.25 mg/kg at the beginning of PCI (Staged-dose PCI Group [0.5+0.25 mg/kg]); while, those have no indication for subsequent PCI will not receive additional anticoagulation (Standard-dose Group [0.5 mg/kg]).
  All patients in the Planned Single-dose Group will receive enoxaparin 0.75 mg/kg at the beginning of coronary angiography no matter they will undergo subsequent PCI (Single-dose PCI Group [0.75 mg/kg]) or not (High-dose Group [0.75 mg/kg]).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enoxaparin (Staged-dose PCI Group) (Experimental): Enoxaparin 0.5 mg/kg at the beginning of coronary angiography (i.e., insertion of angiographic catheter) and additional enoxaparin 0.25 mg/kg at the beginning of PCI (i.e., insertion of guiding catheter).
  Interventions: Drug: Enoxaparin (Staged-dose PCI Group)
- Enoxaparin (Single-dose PCI Group) (Active Comparator): Enoxaparin 0.75 mg/kg at the beginning of coronary angiography (i.e., insertion of angiographic catheter) and NO additional enoxaparin at the beginning of PCI (i.e., insertion of guiding catheter).
  Interventions: Drug: Enoxaparin (Single-dose PCI Group)
- Enoxaparin (High-dose Group) (Experimental): Enoxaparin 0.75 mg/kg at the beginning of coronary angiography (i.e., insertion of angiographic catheter).
  Interventions: Drug: Enoxaparin (High-dose Group)
- Enoxaparin (Standard-dose Group) (Active Comparator): Enoxaparin 0.5 mg/kg at the beginning of coronary angiography (i.e., insertion of angiographic catheter).
  Interventions: Drug: Enoxaparin (Standard-dose Group)

INTERVENTIONS:
Drug: Enoxaparin (Staged-dose PCI Group) — Enoxaparin 0.5+0.25 mg/kg administered intravenously.
  Other Names: Clexane
  Arms: Enoxaparin (Staged-dose PCI Group)
Drug: Enoxaparin (Single-dose PCI Group) — Enoxaparin 0.75 mg/kg administered intravenously.
  Other Names: Clexane
  Arms: Enoxaparin (Single-dose PCI Group)
Drug: Enoxaparin (High-dose Group) — Enoxaparin 0.75 mg/kg administered intravenously.
  Other Names: Clexane
  Arms: Enoxaparin (High-dose Group)
Drug: Enoxaparin (Standard-dose Group) — Enoxaparin 0.5 mg/kg administered intravenously.
  Other Names: Clexane
  Arms: Enoxaparin (Standard-dose Group)

SUMMARY:
The OPTIENOX-PCI is a single-center, prospective, randomized, open-label, controlled study, which is designed to assess the anticoagulation profile of: 1) High-dose (0.75 mg/kg) vs. Standard-dose (0.5 mg/kg) enoxaparin; 2) Staged-dose (0.5+0.25 mg/kg) vs. Single-dose (0.75 mg/kg) enoxaparin in about 376 patients who plan to undergo elective trans-radial coronary angiography (CAG) with or without subsequent percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Once the radial sheaths are successfully inserted, eligible patients will be consecutively, sequentially, and randomly assigned in a 1:1 ratio and with a block size of 4 to either the Planned Single-dose group (0.75 mg/kg) or the Planned Staged-dose group (0.5 ± 0.25 mg/kg).

The first dose enoxaparin will be administered immediately after randomization. In the Planned Single-dose group, enoxaparin 0.75 mg/kg will be given to all patients before CAG irrespective of whether they will undergo subsequent PCI or not. In the Planned Staged-dose group, enoxaparin 0.5 mg/kg will be administered to all patients before CAG and additional 0.25 mg/kg will be given only to those who will undergo subsequent PCI immediately before PCI.

Trans-radial CAG will be performed immediately after the first dose enoxaparin is given. When the angiographic results are available, whether the patients will proceed to subsequent PCI or not will be at the discretion of the procedure operators, who are blinded to the assignment of enoxaparin dosing regimens. Patients who undergo CAG alone in each group will be defined as the High-dose (0.75 mg/kg) and the Standard-dose (0.5 mg/kg) groups, respectively; while, patients who undergo both CAG and subsequent PCI in each group will be defined as the Single-dose PCI (0.75 mg/kg) and the Staged-dose PCI (0.5 + 0.25 mg/kg) groups, respectively.

Anti-Xa levels will be assessed: 1) at 0 min (immediately before), 10 min and 90 min after the first dose enoxaparin is given (CAG-0 min, CAG-10 min, and CAG-90 min, respectively) in all patients; 2) at 0 min (immediately before) and 10 min after the beginning of PCI (PCI-0 min and PCI-10 min, respectively), and at the end of PCI (PCI-End) in patients undergoing PCI.

Target anticoagulation is defined as: 1) anti-Xa level of 0.5-1.8 IU/ml in patients in the High-dose and Standard-dose groups; 2) anti-Xa level of 0.5-1.2 IU/ml before PCI and anti-Xa level of 0.5-1.8 IU/ml from the beginning of PCI up to 90 min after the first dose enoxaparin is given in the Single-dose PCI and the Staged-dose PCI groups.

The information on cardiac ischemic and bleeding events will be collected 24 h after randomization.

The OPTIENOX-PCI study will assess the anticoagulation profile between: 1) the High-dose and the Standard-dose groups (0.75 mg/kg vs. 0.5 mg/kg); 2) the Staged-dose PCI and the Single-dose PCI groups (0.5+0.25 mg/kg vs. 0.75 mg/kg). The result of the present study will provide pharmacodynamical data for the design of future outcome studies.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Aged 18 years or older, male or female.
3. Documented stable coronary artery disease (SCAD) or non-ST-segment elevation acute coronary syndromes (NSTE-ACS).
4. Plan to undergo elective trans-radial coronary angiography with or without subsequent PCI.
5. No fibrinolytic, or anticoagulant, or parenteral antiplatelet therapy within 7 days of screening.
6. Negative cardiac troponin test within 7 days of screening.
7. Trans-radial approach successfully established.
8. Females who are either post-menopausal > 1 year or surgically sterile.

Exclusion Criteria:

1. Recent (within 30 days of screening) acute myocardial infarction, including ST-segment elevation myocardial infarction or non-ST-segment elevation myocardial infarction.
2. The aim of the index coronary angiography is to undergo primary PCI or early PCI for acute coronary syndromes.
3. Any indications other than coronary artery disease (e.g., atrial fibrillation, prosthetic heart valve, venous thromboembolism, ventricular thrombosis, et al) for fibrinolytic or anticoagulant treatment during study period.
4. Planned use of any fibrinolytic or antithrombotic agents, with the exception of enoxaparin, aspirin, clopidogrel, and ticagrelor during study period.
5. Planned coronary artery bypass graft (CABG) during study period.
6. Increased bleeding risk, including

   * any history of intracranial, intraocular, retroperitoneal, or spinal bleeding;
   * recent (within 30 days of screening) gastrointestinal (GI) bleeding;
   * recent (within 30 days of screening) major trauma or major surgery;
   * planned surgery or other invasive procedure during study period;
   * sustained uncontrolled hypertension (systolic blood pressure [SBP] > 180 mmHg or diastolic blood pressure [DBP] > 100 mmHg) within 7 days of screening;
   * history of hemorrhagic disorders, e.g., haemophilia, von Willebrand's disease;
   * inability to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during study period;
   * platelet count less than 100,000/mm3 or hemoglobin < 10 g/dL within 7 days of screening.
7. Contraindications for enoxaparin, e.g., hypersensitivity, active bleeding, bleeding diathesis, coagulation disorders, acute infectious endocarditis, thrombocytopenia (including heparin-induced thrombocytopenia), cerebral hemorrhage, severe liver of kidney diseases, severe hypertension, stroke, retinopathy, et al.
8. History of intolerance to enoxaparin.
9. Patient requires dialysis or has a creatinine clearance < 30 mL/min as calculated by the Cockcroft-Gault equation: Clcr = (140 - Age) × WT / (72 × Scr) (× 0.85 for females), where WT is weight in kg, Scr is serum creatinine in mg/dL measured within 7 days of screening.
10. Any acute or chronic unstable conditions in the past 30 days which, in the opinion of the investigator, may either put the patient at risk or influence the result of the study, e.g., active cancer, et al.
11. Any condition that may increase the risk of non-compliance to study protocol or follow-up, e.g., history of drug addiction or alcohol abuse, et al.
12. Patients who has previously been randomized in this study.
13. Participation in another investigational drug or device study within 30 days of screening.
14. Involvement in the planning and conduct of the study (applies to investigators, contract research organization staff, and study site staff).
15. Known pregnancy, breast-feeding, or intend to become pregnant during the study period.
16. Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Anti-Xa level (CAG-90 min) in the High-dose vs. the Standard-dose group. | At 90 min after the first dose enoxaparin is given.
  The anti-Xa level (CAG-90 min) in the High-dose vs. the Standard-dose group.
Anti-Xa level (CAG-90 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 90 min after the first dose enoxaparin is given.
  The anti-Xa level (CAG-90 min) in the Staged-dose PCI vs. the Single-dose PCI group.

SECONDARY OUTCOMES:
Anti-Xa level (CAG-10 min) in the High-dose vs. the Standard-dose group. | At 10 min after the first dose enoxaparin is given.
  The anti-Xa level (CAG-10 min) in the High-dose vs. the Standard-dose group.
Anti-Xa level (CAG-10 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 10 min after the first dose enoxaparin is given.
  The anti-Xa level (CAG-10 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Anti-Xa level (PCI-0 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 0 min (immediately before) PCI.
  The anti-Xa level (PCI-0 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Anti-Xa level (PCI-10 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 10 min after the beginning of PCI.
  The anti-Xa level (PCI-10 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Anti-Xa level (PCI-End) in the Staged-dose PCI vs. the Single-dose PCI group. | At the end of PCI.
  The anti-Xa level (PCI-End) in the Staged-dose PCI vs. the Single-dose PCI group.
Target anticoagulation (CAG-90 min) in the High-dose vs. the Standard-dose group. | At 90 min after the first dose enoxaparin is given.
  The rate of target anticoagulation (CAG-90 min) in the High-dose vs. the Standard-dose group.
Target anticoagulation (CAG-90 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 90 min after the first dose enoxaparin is given.
  The rate of target anticoagulation (CAG-90 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Target anticoagulation (CAG-10 min) in the High-dose vs. the Standard-dose group. | At 10 min after the first dose enoxaparin is given.
  The rate of target anticoagulation (CAG-10 min) in the High-dose vs. the Standard-dose group.
Target anticoagulation (CAG-10 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 10 min after the first dose enoxaparin is given.
  The rate of target anticoagulation (CAG-10 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Target anticoagulation (PCI-0 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 0 min (immediately before) PCI.
  The rate of target anticoagulation (PCI-0 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Target anticoagulation (PCI-10 min) in the Staged-dose PCI vs. the Single-dose PCI group. | At 10 min after the beginning of PCI.
  The rate of target anticoagulation (PCI-10 min) in the Staged-dose PCI vs. the Single-dose PCI group.
Target anticoagulation (PCI-End) in the Staged-dose PCI vs. the Single-dose PCI group. | At the end of PCI.
  The rate of target anticoagulation (PCI-End) in the Staged-dose PCI vs. the Single-dose PCI group.

OTHER OUTCOMES:
Major adverse cardiac events (MACE) in the High-dose vs. the Standard-dose group. | Up to 24 hours.
  The proportion of patients with the composite of death, or myocardial infarction, or urgent coronary revascularization, or definite or probable stent thrombosis in the High-dose vs. the Standard-dose group.
Major adverse cardiac events (MACE) in the Staged-dose PCI vs. the Single-dose PCI group. | Up to 24 hours.
  The proportion of patients with the composite of death, or myocardial infarction, or urgent coronary revascularization, or definite or probable stent thrombosis in the Staged-dose PCI vs. the Single-dose PCI group.
Thrombolysis in myocardial infarction (TIMI) major or minor bleeding in the High-dose vs. the Standard-dose group. | Up to 24 hours.
  The proportion of patients with the composite of TIMI major or minor bleeding in the High-dose vs. the Standard-dose group.
Thrombolysis in myocardial infarction (TIMI) major or minor bleeding in the Staged-dose PCI vs. the Single-dose PCI group. | Up to 24 hours.
  The proportion of patients with the composite of TIMI major or minor bleeding in the Staged-dose PCI vs. the Single-dose PCI group.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Liu, M.D., Principal Investigator — Department of Cardiology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members; Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):2354-94. doi: 10.1161/CIR.0000000000000133. Epub 2014 Sep 23. No abstract available. PMID 25249586
- [Result] Argenti D, Hoppensteadt D, Heald D, Jensen B, Fareed J. Pharmacokinetics of enoxaparin in patients undergoing percutaneous coronary intervention with and without glycoprotein IIb/IIIa therapy. Am J Ther. 2003 Jul-Aug;10(4):241-6. doi: 10.1097/00045391-200307000-00002. PMID 12845386
- [Result] Bernat I, Horak D, Stasek J, Mates M, Pesek J, Ostadal P, Hrabos V, Dusek J, Koza J, Sembera Z, Brtko M, Aschermann O, Smid M, Polansky P, Al Mawiri A, Vojacek J, Bis J, Costerousse O, Bertrand OF, Rokyta R. ST-segment elevation myocardial infarction treated by radial or femoral approach in a multicenter randomized clinical trial: the STEMI-RADIAL trial. J Am Coll Cardiol. 2014 Mar 18;63(10):964-72. doi: 10.1016/j.jacc.2013.08.1651. Epub 2013 Nov 21. PMID 24211309
- [Result] Caputo RP, Tremmel JA, Rao S, Gilchrist IC, Pyne C, Pancholy S, Frasier D, Gulati R, Skelding K, Bertrand O, Patel T. Transradial arterial access for coronary and peripheral procedures: executive summary by the Transradial Committee of the SCAI. Catheter Cardiovasc Interv. 2011 Nov 15;78(6):823-39. doi: 10.1002/ccd.23052. Epub 2011 May 4. PMID 21544927
- [Result] Chen WH, Lau CP, Lau YK, Ng W, Lee PY, Yu CM, Ma E. Stable and optimal anticoagulation is achieved with a single dose of intravenous enoxaparin in patients undergoing percutaneous coronary intervention. J Invasive Cardiol. 2002 Aug;14(8):439-42. PMID 12147872
- [Result] Chew DP, Bhatt DL, Lincoff AM, Moliterno DJ, Brener SJ, Wolski KE, Topol EJ. Defining the optimal activated clotting time during percutaneous coronary intervention: aggregate results from 6 randomized, controlled trials. Circulation. 2001 Feb 20;103(7):961-6. doi: 10.1161/01.cir.103.7.961. PMID 11181470
- [Result] Choussat R, Montalescot G, Collet JP, Vicaut E, Ankri A, Gallois V, Drobinski G, Sotirov I, Thomas D. A unique, low dose of intravenous enoxaparin in elective percutaneous coronary intervention. J Am Coll Cardiol. 2002 Dec 4;40(11):1943-50. doi: 10.1016/s0735-1097(02)02531-7. PMID 12475453
- [Result] Cohen M. The role of low-molecular-weight heparin in the management of acute coronary syndromes. J Am Coll Cardiol. 2003 Feb 19;41(4 Suppl S):55S-61S. doi: 10.1016/s0735-1097(02)02901-7. PMID 12644342
- [Result] Collet JP, Montalescot G, Lison L, Choussat R, Ankri A, Drobinski G, Sotirov I, Thomas D. Percutaneous coronary intervention after subcutaneous enoxaparin pretreatment in patients with unstable angina pectoris. Circulation. 2001 Feb 6;103(5):658-63. doi: 10.1161/01.cir.103.5.658. PMID 11156876
- [Result] Feldman DN, Swaminathan RV, Kaltenbach LA, Baklanov DV, Kim LK, Wong SC, Minutello RM, Messenger JC, Moussa I, Garratt KN, Piana RN, Hillegass WB, Cohen MG, Gilchrist IC, Rao SV. Adoption of radial access and comparison of outcomes to femoral access in percutaneous coronary intervention: an updated report from the national cardiovascular data registry (2007-2012). Circulation. 2013 Jun 11;127(23):2295-306. doi: 10.1161/CIRCULATIONAHA.112.000536. PMID 23753843
- [Result] Ferguson JJ, Dougherty KG, Gaos CM, Bush HS, Marsh KC, Leachman DR. Relation between procedural activated coagulation time and outcome after percutaneous transluminal coronary angioplasty. J Am Coll Cardiol. 1994 Apr;23(5):1061-5. doi: 10.1016/0735-1097(94)90590-8. PMID 8144768
- [Result] Ferrante G, Rao SV, Juni P, Da Costa BR, Reimers B, Condorelli G, Anzuini A, Jolly SS, Bertrand OF, Krucoff MW, Windecker S, Valgimigli M. Radial Versus Femoral Access for Coronary Interventions Across the Entire Spectrum of Patients With Coronary Artery Disease: A Meta-Analysis of Randomized Trials. JACC Cardiovasc Interv. 2016 Jul 25;9(14):1419-34. doi: 10.1016/j.jcin.2016.04.014. Epub 2016 Jun 29. PMID 27372195
- [Result] Giugliano RP, White JA, Bode C, Armstrong PW, Montalescot G, Lewis BS, van 't Hof A, Berdan LG, Lee KL, Strony JT, Hildemann S, Veltri E, Van de Werf F, Braunwald E, Harrington RA, Califf RM, Newby LK; EARLY ACS Investigators. Early versus delayed, provisional eptifibatide in acute coronary syndromes. N Engl J Med. 2009 May 21;360(21):2176-90. doi: 10.1056/NEJMoa0901316. Epub 2009 Mar 30. PMID 19332455
- [Result] Gurm HS, Hosman C, Share D, Moscucci M, Hansen BB; Blue Cross Blue Shield of Michigan Cardiovascular Consortium. Comparative safety of vascular closure devices and manual closure among patients having percutaneous coronary intervention. Ann Intern Med. 2013 Nov 19;159(10):660-6. doi: 10.7326/0003-4819-159-10-201311190-00004. PMID 24247671
- [Result] Hirsh J, Raschke R. Heparin and low-molecular-weight heparin: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):188S-203S. doi: 10.1378/chest.126.3_suppl.188S. PMID 15383472
- [Result] Karrowni W, Vyas A, Giacomino B, Schweizer M, Blevins A, Girotra S, Horwitz PA. Radial versus femoral access for primary percutaneous interventions in ST-segment elevation myocardial infarction patients: a meta-analysis of randomized controlled trials. JACC Cardiovasc Interv. 2013 Aug;6(8):814-23. doi: 10.1016/j.jcin.2013.04.010. PMID 23968700
- [Result] Kereiakes DJ, Grines C, Fry E, Esente P, Hoppensteadt D, Midei M, Barr L, Matthai W, Todd M, Broderick T, Rubinstein R, Fareed J, Santoian E, Neiderman A, Brodie B, Zidar J, Ferguson JJ, Cohen M; NICE 1 and NICE 4 Investigators. National Investigators Collaborating on Enoxaparin. Enoxaparin and abciximab adjunctive pharmacotherapy during percutaneous coronary intervention. J Invasive Cardiol. 2001 Apr;13(4):272-8. PMID 11287711
- [Result] Kerre S, Kustermans L, Vandendriessche T, Bosmans J, Haine SE, Miljoen H, Vrints CJ, Beutels P, Wouters K, Claeys MJ. Cost-effectiveness of contemporary vascular closure devices for the prevention of vascular complications after percutaneous coronary interventions in an all-comers PCI population. EuroIntervention. 2014 Jun;10(2):191-7. doi: 10.4244/EIJV10I2A32. PMID 24952056
- [Result] Khambatta S, Othman H, Seth M, Lalonde T, Rosman HS, Gurm HS, Mehta RH; Blue Cross Blue Shield of Michigan Cardiovascular Consortium (BMC2) Investigators. Association Of Bleeding Avoidance Strategies with age-related bleeding and In-hospital mortality in patients undergoing percutaneous coronary Interventions. Cardiovasc Revasc Med. 2016 Jun;17(4):233-40. doi: 10.1016/j.carrev.2016.02.014. Epub 2016 Feb 27. PMID 26994504
- [Result] Lee MS, Applegate B, Rao SV, Kirtane AJ, Seto A, Stone GW. Minimizing femoral artery access complications during percutaneous coronary intervention: a comprehensive review. Catheter Cardiovasc Interv. 2014 Jul 1;84(1):62-9. doi: 10.1002/ccd.25435. Epub 2014 Mar 10. PMID 24677734
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Result] Martin JL, Fry ET, Sanderink GJ, Atherley TH, Guimart CM, Chevalier PJ, Ozoux ML, Pensyl CE, Bigonzi F. Reliable anticoagulation with enoxaparin in patients undergoing percutaneous coronary intervention: The pharmacokinetics of enoxaparin in PCI (PEPCI) study. Catheter Cardiovasc Interv. 2004 Feb;61(2):163-70. doi: 10.1002/ccd.10726. PMID 14755805
- [Result] Mauri L, Hsieh WH, Massaro JM, Ho KK, D'Agostino R, Cutlip DE. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med. 2007 Mar 8;356(10):1020-9. doi: 10.1056/NEJMoa067731. Epub 2007 Feb 12. PMID 17296821
- [Result] McGarry TF Jr, Gottlieb RS, Morganroth J, Zelenkofske SL, Kasparian H, Duca PR, Lester RM, Kreulen TH. The relationship of anticoagulation level and complications after successful percutaneous transluminal coronary angioplasty. Am Heart J. 1992 Jun;123(6):1445-51. doi: 10.1016/0002-8703(92)90793-u. PMID 1595522
- [Result] Montalescot G, Collet JP, Tanguy ML, Ankri A, Payot L, Dumaine R, Choussat R, Beygui F, Gallois V, Thomas D. Anti-Xa activity relates to survival and efficacy in unselected acute coronary syndrome patients treated with enoxaparin. Circulation. 2004 Jul 27;110(4):392-8. doi: 10.1161/01.CIR.0000136830.65073.C7. Epub 2004 Jul 12. PMID 15249498
- [Result] Montalescot G, White HD, Gallo R, Cohen M, Steg PG, Aylward PE, Bode C, Chiariello M, King SB 3rd, Harrington RA, Desmet WJ, Macaya C, Steinhubl SR; STEEPLE Investigators. Enoxaparin versus unfractionated heparin in elective percutaneous coronary intervention. N Engl J Med. 2006 Sep 7;355(10):1006-17. doi: 10.1056/NEJMoa052711. PMID 16957147
- [Result] Montalescot G, Cohen M, Salette G, Desmet WJ, Macaya C, Aylward PE, Steg PG, White HD, Gallo R, Steinhubl SR; STEEPLE Investigators. Impact of anticoagulation levels on outcomes in patients undergoing elective percutaneous coronary intervention: insights from the STEEPLE trial. Eur Heart J. 2008 Feb;29(4):462-71. doi: 10.1093/eurheartj/ehn008. PMID 18276619
- [Result] Montalescot G, Zeymer U, Silvain J, Boulanger B, Cohen M, Goldstein P, Ecollan P, Combes X, Huber K, Pollack C Jr, Benezet JF, Stibbe O, Filippi E, Teiger E, Cayla G, Elhadad S, Adnet F, Chouihed T, Gallula S, Greffet A, Aout M, Collet JP, Vicaut E; ATOLL Investigators. Intravenous enoxaparin or unfractionated heparin in primary percutaneous coronary intervention for ST-elevation myocardial infarction: the international randomised open-label ATOLL trial. Lancet. 2011 Aug 20;378(9792):693-703. doi: 10.1016/S0140-6736(11)60876-3. PMID 21856483
- [Result] Narins CR, Hillegass WB Jr, Nelson CL, Tcheng JE, Harrington RA, Phillips HR, Stack RS, Califf RM. Relation between activated clotting time during angioplasty and abrupt closure. Circulation. 1996 Feb 15;93(4):667-71. doi: 10.1161/01.cir.93.4.667. PMID 8640994
- [Result] Navarese EP, De Luca G, Castriota F, Kozinski M, Gurbel PA, Gibson CM, Andreotti F, Buffon A, Siller-Matula JM, Sukiennik A, De Servi S, Kubica J. Low-molecular-weight heparins vs. unfractionated heparin in the setting of percutaneous coronary intervention for ST-elevation myocardial infarction: a meta-analysis. J Thromb Haemost. 2011 Oct;9(10):1902-15. doi: 10.1111/j.1538-7836.2011.04445.x. PMID 21777368
- [Result] Rao SV, Ou FS, Wang TY, Roe MT, Brindis R, Rumsfeld JS, Peterson ED. Trends in the prevalence and outcomes of radial and femoral approaches to percutaneous coronary intervention: a report from the National Cardiovascular Data Registry. JACC Cardiovasc Interv. 2008 Aug;1(4):379-86. doi: 10.1016/j.jcin.2008.05.007. PMID 19463333
- [Result] Rao SV, Cohen MG, Kandzari DE, Bertrand OF, Gilchrist IC. The transradial approach to percutaneous coronary intervention: historical perspective, current concepts, and future directions. J Am Coll Cardiol. 2010 May 18;55(20):2187-95. doi: 10.1016/j.jacc.2010.01.039. PMID 20466199
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Result] Sachdeva S, Saha S. Transradial approach to cardiovascular interventions: an update. Int J Angiol. 2014 Jun;23(2):77-84. doi: 10.1055/s-0034-1372243. PMID 25075159
- [Result] Samama MM, Gerotziafas GT. Comparative pharmacokinetics of LMWHs. Semin Thromb Hemost. 2000;26 Suppl 1:31-8. doi: 10.1055/s-2000-9497. PMID 11011804
- [Result] Sanborn TA, Tomey MI, Mehran R, Genereux P, Witzenbichler B, Brener SJ, Kirtane AJ, McAndrew TC, Kornowski R, Dudek D, Nikolsky E, Stone GW. Femoral vascular closure device use, bivalirudin anticoagulation, and bleeding after primary angioplasty for STEMI: results from the HORIZONS-AMI trial. Catheter Cardiovasc Interv. 2015 Feb 15;85(3):371-9. doi: 10.1002/ccd.25663. Epub 2014 Oct 28. PMID 25179260
- [Result] Sanchez-Pena P, Hulot JS, Urien S, Ankri A, Collet JP, Choussat R, Lechat P, Montalescot G. Anti-factor Xa kinetics after intravenous enoxaparin in patients undergoing percutaneous coronary intervention: a population model analysis. Br J Clin Pharmacol. 2005 Oct;60(4):364-73. doi: 10.1111/j.1365-2125.2005.02452.x. PMID 16187968
- [Result] Silvain J, Beygui F, Ankri A, Bellemain-Appaix A, Pena A, Barthelemy O, Cayla G, Gallois V, Galier S, Costagliola D, Collet JP, Montalescot G. Enoxaparin anticoagulation monitoring in the catheterization laboratory using a new bedside test. J Am Coll Cardiol. 2010 Feb 16;55(7):617-25. doi: 10.1016/j.jacc.2009.08.077. PMID 20170785
- [Result] Silvain J, Beygui F, Barthelemy O, Pollack C Jr, Cohen M, Zeymer U, Huber K, Goldstein P, Cayla G, Collet JP, Vicaut E, Montalescot G. Efficacy and safety of enoxaparin versus unfractionated heparin during percutaneous coronary intervention: systematic review and meta-analysis. BMJ. 2012 Feb 3;344:e553. doi: 10.1136/bmj.e553. PMID 22306479
- [Result] Stone GW, White HD, Ohman EM, Bertrand ME, Lincoff AM, McLaurin BT, Cox DA, Pocock SJ, Ware JH, Feit F, Colombo A, Manoukian SV, Lansky AJ, Mehran R, Moses JW; Acute Catheterization and Urgent Intervention Triage strategy (ACUITY) trial investigators. Bivalirudin in patients with acute coronary syndromes undergoing percutaneous coronary intervention: a subgroup analysis from the Acute Catheterization and Urgent Intervention Triage strategy (ACUITY) trial. Lancet. 2007 Mar 17;369(9565):907-19. doi: 10.1016/S0140-6736(07)60450-4. PMID 17368152
- [Result] Dose-ranging trial of enoxaparin for unstable angina: results of TIMI 11A. The Thrombolysis in Myocardial Infarction (TIMI) 11A Trial Investigators. J Am Coll Cardiol. 1997 Jun;29(7):1474-82. PMID 9180107
- [Result] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Result] Tolleson TR, O'Shea JC, Bittl JA, Hillegass WB, Williams KA, Levine G, Harrington RA, Tcheng JE. Relationship between heparin anticoagulation and clinical outcomes in coronary stent intervention: observations from the ESPRIT trial. J Am Coll Cardiol. 2003 Feb 5;41(3):386-93. doi: 10.1016/s0735-1097(02)02767-5. PMID 12575964
- [Result] Valgimigli M, Gagnor A, Calabro P, Frigoli E, Leonardi S, Zaro T, Rubartelli P, Briguori C, Ando G, Repetto A, Limbruno U, Cortese B, Sganzerla P, Lupi A, Galli M, Colangelo S, Ierna S, Ausiello A, Presbitero P, Sardella G, Varbella F, Esposito G, Santarelli A, Tresoldi S, Nazzaro M, Zingarelli A, de Cesare N, Rigattieri S, Tosi P, Palmieri C, Brugaletta S, Rao SV, Heg D, Rothenbuhler M, Vranckx P, Juni P; MATRIX Investigators. Radial versus femoral access in patients with acute coronary syndromes undergoing invasive management: a randomised multicentre trial. Lancet. 2015 Jun 20;385(9986):2465-76. doi: 10.1016/S0140-6736(15)60292-6. Epub 2015 Mar 16. PMID 25791214
- [Result] Wimmer NJ, Secemsky EA, Mauri L, Roe MT, Saha-Chaudhuri P, Dai D, McCabe JM, Resnic FS, Gurm HS, Yeh RW. Effectiveness of Arterial Closure Devices for Preventing Complications With Percutaneous Coronary Intervention: An Instrumental Variable Analysis. Circ Cardiovasc Interv. 2016 Apr;9(4):e003464. doi: 10.1161/CIRCINTERVENTIONS.115.003464. PMID 27059685
- [Result] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339